CLINICAL TRIAL: NCT06724770
Title: Diseño De Una Intervención Para Dotar a Mandos Intermedios Y Directivos De Instituciones Sanitarias Con Herramientas Para Incrementar La Resiliencia De Sus Equipos
Brief Title: Design of an Intervention to Equip Middle Managers and Managers in Healthcare Institutions with Tools to Increase the Resilience of Their Teams
Acronym: e-Resiliencia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Irene Carrillo Murcia (Other)
Collaborators: Foundation for the Promotion of Healthcare and Biomedical Research in the Valencian Community (FISABIO) (Unknown)
Responsible Party: Sponsor-Investigator, Irene Carrillo Murcia, Assistant Professor, Universidad Miguel Hernandez de Elche
Organization: Universidad Miguel Hernandez de Elche (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ILISABIO22_AP09
Record Dates: First submitted 2024-11-29; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Occupational Health; Resilience; Job Stress; Well-being At Work; Highly Stressful Situations; Healthcare Worker
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Intervention Model Description: Participants voluntarily adhere to the intervention. The intervention consists of the review and use of the e-Resilience tool. It is a toolkit that provides training in skills to strengthen the resilience of teams working in healthcare institutions. Participants complete knowledge questionnaires before and after the intervention. There is no control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- e-Resilience Intervention (Experimental): Middle management and healthcare professionals who voluntarily participate in the e-Resilience intervention.
  Interventions: Other: Resilience training intervention

INTERVENTIONS:
Other: Resilience training intervention — Training intervention on tools and strategies to strengthen the resilience of work teams in healthcare centres.

SUMMARY:
The main objective of this preparatory action (experimental study without control group, before and after measurements) is to develop and test the feasibility of the e-Resilience tool in a relevant environment (TRL6). This web-based tool has been designed to facilitate the work of the top and middle management of healthcare institutions to strengthen the resilience of their teams to face critical situations inherent to healthcare activity.

The main questions it aims to answer are:

1. Which components of the e-Resilience intervention need to be improved?
2. Does the e-Resilience tool improve the knowledge of middle managers in healthcare institutions on specific techniques and strategies to strengthen the resilience of the professionals and teams under their care?
3. Is the e-Resilience tool helpful and applicable to clinical settings in the opinion of middle managers in healthcare institutions?

Participants in the study are middle management and healthcare professionals from primary care centres and hospitals in the Valencian Community (Spain). A group of experts review the components of the intervention/tool to improve its adaptability to clinical settings. Subsequently, a sample of healthcare professionals and middle managers complete the intervention by answering a knowledge questionnaire before and after the intervention and a survey to evaluate the tool.

There is no control group.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals and middle management in active healthcare institutions.

Exclusion Criteria:

* Inability to complete the web-based intervention due to access difficulties or lack of digital literacy.

Ages: 26 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Number of incorporations and adaptations necessary for the validation of e-Resilience in a relevant environment. | 5 months
  Number of change proposals of the expert group to adapt the tool to the target environments' needs and enhance its applicability.
Hits on resilience knowledge questionnaire (pre-intervention). | 3 months
  Number of correct answers to questions on knowledge of models, techniques, tools and strategies for building resilience in clinical settings.
Hits on resilience knowledge questionnaire (post-intervention). | 3 months
  Number of correct answers to questions on knowledge of models, techniques, tools and strategies for building resilience in clinical settings.

SECONDARY OUTCOMES:
Clarity of the e-Resilience tool components. | 3 months
  Clarity of the e-Resilience tool components (scale 1-5, where 1 = not clear at all and 5 = totally clear).
Usefulness and applicability of the e-Resilience tool. | 3 months
  Usefulness and applicability of the e-Resilience tool (scale 1-5, where 1 = not useful or applicable at all and 5 = fully useful and applicable).
Perception of improvement of own capacity to strengthen the resilience of healthcare teams. | 3 months
  The contents of the course have allowed me to learn strategies to strengthen the resilience of the professionals or teams in my charge (scale 1-5, where 1 = strongly disagree and 5 = strongly agree).
Willingness to recommend e-Resilience. | 3 months
  I will recommend the intervention to other colleagues (scale 1-5, where 1 = strongly disagree and 5 = strongly agree).
Willingness to use e-Resilience in the future. | 3 months
  I will apply any of the tools or strategies learned to strengthen individual, team or organisational resilience in my work environment. (scale 1-5, where 1 = strongly disagree and 5 = strongly agree).
Overall satisfaction with the e-Resilience intervention. | 3 months
  Overall satisfaction with the e-Resilience intervention (scale 0-10, where 0 = not at all satisfied and 10 = completely satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Miguel Hernández de Elche, Elche, Alicante, Spain

REFERENCES:
- [Background] Seys D, Panella M, Russotto S, Strametz R, Joaquin Mira J, Van Wilder A, Godderis L, Vanhaecht K. In search of an international multidimensional action plan for second victim support: a narrative review. BMC Health Serv Res. 2023 Jul 31;23(1):816. doi: 10.1186/s12913-023-09637-8. PMID 37525127
- [Background] Mira JJ, Vicente MA, Lopez-Pineda A, Carrillo I, Guilabert M, Fernandez C, Perez-Jover V, Martin Delgado J, Perez-Perez P, Cobos Vargas A, Astier-Pena MP, Martinez-Garcia OB, Marco-Gomez B, Abad Bouzan C. Preventing and Addressing the Stress Reactions of Health Care Workers Caring for Patients With COVID-19: Development of a Digital Platform (Be + Against COVID). JMIR Mhealth Uhealth. 2020 Oct 5;8(10):e21692. doi: 10.2196/21692. PMID 32936769
- [Background] Venegas CL, Nkangu MN, Duffy MC, Fergusson DA, Spilg EG. Interventions to improve resilience in physicians who have completed training: A systematic review. PLoS One. 2019 Jan 17;14(1):e0210512. doi: 10.1371/journal.pone.0210512. eCollection 2019. PMID 30653550
- [Background] Stoliker BE, Vaughan AD, Collins J, Black M, Anderson GS. Building Personal Resilience following an Online Resilience Training Program for BScN Students. West J Nurs Res. 2022 Aug;44(8):755-764. doi: 10.1177/01939459211017240. Epub 2021 May 17. PMID 33998338
- [Background] Strametz R, Raspe M, Ettl B, Huf W, Pitz A. [Recommended actions: Reinforcing clinicians' resilience and supporting second victims during the COVID-19 pandemic to maintain capacity in the healthcare system]. Zentralbl Arbeitsmed Arbeitsschutz Ergon. 2020;70(6):264-268. doi: 10.1007/s40664-020-00405-7. Epub 2020 Sep 2. German. PMID 32905028
- [Background] Raetze S, Duchek S, Maynard MT, Wohlgemuth M. Resilience in organization-related research: An integrative conceptual review across disciplines and levels of analysis. J Appl Psychol. 2022 Jun;107(6):867-897. doi: 10.1037/apl0000952. Epub 2021 Nov 11. PMID 34766796
- [Background] Daly LM. Resilience: An Integrated Review. Nurs Sci Q. 2020 Oct;33(4):330-338. doi: 10.1177/0894318420943141. PMID 32940160
- [Background] Winwood PC, Colon R, McEwen K. A practical measure of workplace resilience: developing the resilience at work scale. J Occup Environ Med. 2013 Oct;55(10):1205-12. doi: 10.1097/JOM.0b013e3182a2a60a. PMID 24064782
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Wagnild GM, Young HM. Development and psychometric evaluation of the Resilience Scale. J Nurs Meas. 1993 Winter;1(2):165-78. PMID 7850498
- [Background] Bartone PT, Ursano RJ, Wright KM, Ingraham LH. The impact of a military air disaster on the health of assistance workers. A prospective study. J Nerv Ment Dis. 1989 Jun;177(6):317-28. doi: 10.1097/00005053-198906000-00001. PMID 2723619
- [Background] Wiig S, Aase K, Billett S, Canfield C, Roise O, Nja O, Guise V, Haraldseid-Driftland C, Ree E, Anderson JE, Macrae C; RiH-team. Defining the boundaries and operational concepts of resilience in the resilience in healthcare research program. BMC Health Serv Res. 2020 Apr 19;20(1):330. doi: 10.1186/s12913-020-05224-3. PMID 32306981
- [Background] Sisto A, Vicinanza F, Campanozzi LL, Ricci G, Tartaglini D, Tambone V. Towards a Transversal Definition of Psychological Resilience: A Literature Review. Medicina (Kaunas). 2019 Nov 16;55(11):745. doi: 10.3390/medicina55110745. PMID 31744109
- [Background] Bodenheimer T, Sinsky C. From triple to quadruple aim: care of the patient requires care of the provider. Ann Fam Med. 2014 Nov-Dec;12(6):573-6. doi: 10.1370/afm.1713. PMID 25384822
- [Background] Schwappach DL, Boluarte TA. The emotional impact of medical error involvement on physicians: a call for leadership and organisational accountability. Swiss Med Wkly. 2009 Jan 10;139(1-2):9-15. doi: 10.4414/smw.2009.12417. PMID 18951201
- [Background] Bourne T, Shah H, Falconieri N, Timmerman D, Lees C, Wright A, Lumsden MA, Regan L, Van Calster B. Burnout, well-being and defensive medical practice among obstetricians and gynaecologists in the UK: cross-sectional survey study. BMJ Open. 2019 Nov 25;9(11):e030968. doi: 10.1136/bmjopen-2019-030968. PMID 31767585
- [Background] Schiess C, Schwappach D, Schwendimann R, Vanhaecht K, Burgstaller M, Senn B. A Transactional "Second-Victim" Model-Experiences of Affected Healthcare Professionals in Acute-Somatic Inpatient Settings: A Qualitative Metasynthesis. J Patient Saf. 2021 Dec 1;17(8):e1001-e1018. doi: 10.1097/PTS.0000000000000461. PMID 29384831
- [Background] Sovold LE, Naslund JA, Kousoulis AA, Saxena S, Qoronfleh MW, Grobler C, Munter L. Prioritizing the Mental Health and Well-Being of Healthcare Workers: An Urgent Global Public Health Priority. Front Public Health. 2021 May 7;9:679397. doi: 10.3389/fpubh.2021.679397. eCollection 2021. PMID 34026720
- [Background] Jacobs B, McGovern J, Heinmiller J, Drenkard K. Engaging Employees in Well-Being: Moving From the Triple Aim to the Quadruple Aim. Nurs Adm Q. 2018 Jul/Sep;42(3):231-245. doi: 10.1097/NAQ.0000000000000303. PMID 29870489
- See also: Related Info — https://www.eresiliencia.es/